CLINICAL TRIAL: NCT02457299
Title: A Multicenter, Randomized Trial of Esophagectomy and Cervical Esophagogastrostomy With (Two-stage) or Without (One-stage) Prior Ischemic Gastric Preconditioning by Laparoscopic Ligation of Left Gastric and Short Gastric Arteries
Brief Title: Esophagectomy With or Without Prior Ischemic Gastric Preconditioning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Standard of care was modified at the primary institution
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH15-175
Record Dates: First submitted 2015-04-21; First posted 2015-05-29 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Esophageal Cancer
Keywords: Esophagectomy; Gastric Conduit; Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two Stage Esophagectomy (Active Comparator): Ischemic gastric preconditioning performed 7-10 prior to esophagectomy
  Interventions: Procedure: Two Stage Esophagectomy
- One Stage Esophagectomy (Active Comparator): Esophagectomy alone
  Interventions: Procedure: One Stage Esophagectomy

INTERVENTIONS:
Procedure: Two Stage Esophagectomy — Patients will undergo laparoscopic staging and ischemic gastric conditioning and pyloric Botox injection 7-10 days prior to an esophagectomy with gastric pull-up reconstruction
  Arms: Two Stage Esophagectomy
Procedure: One Stage Esophagectomy — Patients will undergo an esophagectomy with gastric pull-up reconstruction without any preconditioning.
  Arms: One Stage Esophagectomy

SUMMARY:
This multi-center, randomized prospective clinical trial involves esophageal cancer patients who are surgical candidates. Patients will be randomized either to the one stage or the two stage esophagectomy procedure. Surgical, oncology outcomes, quality of life and cost analysis from both types of procedure will be reviewed and compared.

DETAILED DESCRIPTION:
Esophagectomy with gastric pull-up reconstruction is the current preferred operation for either benign or malignant esophageal disease requiring resection. One of the major complications of an esophagectomy with gastric pull-up reconstruction is esophagus-stomach connection (gastric conduit) failure, which carries significant morbidity and mortality. Many factors contribute to the development of gastric conduit failure, but relative decreased blood flow (ischemia) of the tip of the gastric conduit is believed to be one major factor. This is due to the sacrifice of 3 of the 5 gastric blood supplies leaving the tip of the conduit to rely on collateral vessels. In an effort to improve perfusion to the gastric conduit and to minimize ischemia, the relatively novel approach of ischemic gastric preconditioning was devised, but without concrete evidence to show an advantage of a reduction in gastric conduit failures.

Patients meeting eligibility criteria and agree to participation in the study will be randomized to either a esophagectomy with (two-stage) or without (one-stage) ischemic gastric preconditioning and the incidence of gastric conduit failure will be compared. Those randomized to a two-stage procedure will have laparoscopic staging and ischemic gastric conditioning and pyloric Botox injection done 7-10 days prior to an esophagectomy and those randomized to a one-stage procedure will only have the esophagectomy performed.

Validated quality of life (QOL) questionnaires will be completed at the preoperative visit as well as on the day of discharge and at postoperative follow-up timepoints: 3 weeks, 3 months, 6 months, 12 months and 24 months. Data collection will be mostly collected through electronic medical record review and will include, but is not limited to: demographic data; imaging and laboratory values; past medical, surgical and social history; inpatient and intraoperative data; and vitals signs. Patients will be assessed for adverse events throughout study participation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide written informed consent
* Subject is a candidate for esophagectomy with or without gastric pre-conditioning procedure per thoracic surgeon
* Patient is at least 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Cancer stage: T1-2-3 N0M0, Locally advanced, T2-3 N1M0 based on American Joint Committee on Cancer (AJCC) 7th Edition by the oncologist
* No definitive radiological evidence of distant metastases as evaluated by CT or PET/CT scan
* Subject is willing and able to comply with the study procedures and complete the entire study as specified in the protocol, including follow-up visits.

Exclusion Criteria:

* Patients < 18 years old
* History of invasive cancer within the past 5 years, (exceptions: non melanoma skin cancer, in situ cancers)
* Prior upper abdominal surgeries performed open and/or laparoscopic; such as but not limited to Nissen fundoplication, gastrectomy, bariatric surgery, hiatus hernia repair.
* Subject is participating in another investigational trial
* Subject is pregnant or has plans to become pregnant during the study period or is currently breastfeeding
* Subject is part of the site personnel directly involved with this study
* Subject is a family member of the investigational study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The number of participants with gastric conduit failures as a measure of safety and tolerability in the one-stage esophagectomy as compared with the two-stage esophagectomy. | 7-10 days

SECONDARY OUTCOMES:
Mortality rates in both groups | 30-90 days
Cost effectiveness analysis of treatment in one-stage versus two-stage esophagectomy | Hospital inpatient stay, an expected average of a week
Nutritional status of one-stage versus two-stage esophagectomy | Within 30-days of surgery as compared with 3 and 12 month follow-up time points
  This will be determined by prealbumin and albumin values
Quality of Life (QOL) scores of patients in both arms | baseline and up to 24 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ki Wan Kim, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wormuth JK, Heitmiller RF. Esophageal conduit necrosis. Thorac Surg Clin. 2006 Feb;16(1):11-22. doi: 10.1016/j.thorsurg.2006.01.003. PMID 16696279
- [Background] Honkoop P, Siersema PD, Tilanus HW, Stassen LP, Hop WC, van Blankenstein M. Benign anastomotic strictures after transhiatal esophagectomy and cervical esophagogastrostomy: risk factors and management. J Thorac Cardiovasc Surg. 1996 Jun;111(6):1141-6; discussion 1147-8. doi: 10.1016/s0022-5223(96)70215-5. PMID 8642814
- [Background] Cooke DT, Lin GC, Lau CL, Zhang L, Si MS, Lee J, Chang AC, Pickens A, Orringer MB. Analysis of cervical esophagogastric anastomotic leaks after transhiatal esophagectomy: risk factors, presentation, and detection. Ann Thorac Surg. 2009 Jul;88(1):177-84; discussion 184-5. doi: 10.1016/j.athoracsur.2009.03.035. PMID 19559221
- [Background] Yetasook AK, Leung D, Howington JA, Talamonti MS, Zhao J, Carbray JM, Ujiki MB. Laparoscopic ischemic conditioning of the stomach prior to esophagectomy. Dis Esophagus. 2013 Jul;26(5):479-86. doi: 10.1111/j.1442-2050.2012.01374.x. Epub 2012 Jul 20. PMID 22816598
- [Background] Urschel JD. Ischemic conditioning of the rat stomach: implications for esophageal replacement with stomach. J Cardiovasc Surg (Torino). 1995 Apr;36(2):191-3. PMID 7790342
- [Background] Reavis KM, Chang EY, Hunter JG, Jobe BA. Utilization of the delay phenomenon improves blood flow and reduces collagen deposition in esophagogastric anastomoses. Ann Surg. 2005 May;241(5):736-45; discussion 745-7. doi: 10.1097/01.sla.0000160704.50657.32. PMID 15849509
- [Background] Cuenca-Abente F, Assalia A, del Genio G, Rogula T, Nocca D, Ueda K, Gagner M. Laparoscopic partial gastric transection and devascularization in order to enhance its flow. Ann Surg Innov Res. 2008 Jul 7;2:3. doi: 10.1186/1750-1164-2-3. PMID 18606017
- [Background] Akiyama S, Kodera Y, Sekiguchi H, Kasai Y, Kondo K, Ito K, Takagi H. Preoperative embolization therapy for esophageal operation. J Surg Oncol. 1998 Dec;69(4):219-23. doi: 10.1002/(sici)1096-9098(199812)69:43.0.co;2-7. PMID 9881938
- [Background] Bludau M, Holscher AH, Vallbohmer D, Gutschow C, Schroder W. Ischemic conditioning of the gastric conduit prior to esophagectomy improves mucosal oxygen saturation. Ann Thorac Surg. 2010 Oct;90(4):1121-6. doi: 10.1016/j.athoracsur.2010.06.003. PMID 20868800
- [Background] Oezcelik A, Banki F, DeMeester SR, Leers JM, Ayazi S, Abate E, Hagen JA, Lipham JC, DeMeester TR. Delayed esophagogastrostomy: a safe strategy for management of patients with ischemic gastric conduit at time of esophagectomy. J Am Coll Surg. 2009 Jun;208(6):1030-4. doi: 10.1016/j.jamcollsurg.2009.02.055. Epub 2009 Apr 24. PMID 19476888
- [Background] Holscher AH, Schneider PM, Gutschow C, Schroder W. Laparoscopic ischemic conditioning of the stomach for esophageal replacement. Ann Surg. 2007 Feb;245(2):241-6. doi: 10.1097/01.sla.0000245847.40779.10. PMID 17245177
- [Background] Nguyen NT, Longoria M, Sabio A, Chalifoux S, Lee J, Chang K, Wilson SE. Preoperative laparoscopic ligation of the left gastric vessels in preparation for esophagectomy. Ann Thorac Surg. 2006 Jun;81(6):2318-20. doi: 10.1016/j.athoracsur.2005.05.033. PMID 16731189
- [Background] Schroder W, Holscher AH, Bludau M, Vallbohmer D, Bollschweiler E, Gutschow C. Ivor-Lewis esophagectomy with and without laparoscopic conditioning of the gastric conduit. World J Surg. 2010 Apr;34(4):738-43. doi: 10.1007/s00268-010-0403-x. PMID 20098986
- [Background] Sepesi B, Swisher SG, Walsh GL, Correa A, Mehran RJ, Rice D, Roth J, Vaporciyan A, Hofstetter WL. Omental reinforcement of the thoracic esophagogastric anastomosis: an analysis of leak and reintervention rates in patients undergoing planned and salvage esophagectomy. J Thorac Cardiovasc Surg. 2012 Nov;144(5):1146-50. doi: 10.1016/j.jtcvs.2012.07.085. Epub 2012 Aug 28. PMID 22939861
- [Background] Varela E, Reavis KM, Hinojosa MW, Nguyen N. Laparoscopic gastric ischemic conditioning prior to esophagogastrectomy: technique and review. Surg Innov. 2008 Jun;15(2):132-5. doi: 10.1177/1553350608317352. Epub 2008 May 13. PMID 18480085